CLINICAL TRIAL: NCT06761521
Title: Monitoring of Implant Diseases: Diagnosis and Monitoring with AMMP-8 Test Technology: a 5-year Follow-up Study
Brief Title: Monitoring of Implant Diseases: Diagnosis and Monitoring with AMMP-8 Test Technology
Acronym: IMP_TRE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hanna Lahteenmaki (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Hanna Lahteenmaki, Doctor, Dental hygienist, Lahanna oy
Organization: Lahanna oy (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20092024
Record Dates: First submitted 2024-09-25; First posted 2025-01-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implant Health; Peri-Implantitis and Peri-implant Mucositis
Keywords: Ammp-8; Peri-implant diseases; mucositis; prevention; maintenance
MeSH Terms: conditions — Peri-Implantitis; Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients who had participated in a previous study (Other): Bleeding on probing, Peri-implant pocket depth, x-ray findings and aMMP-8 tests will be taking.
  Interventions: Diagnostic Test: Peri-Implantitis and Peri-implant mucositis

INTERVENTIONS:
Diagnostic Test: Peri-Implantitis and Peri-implant mucositis — peri-implant mucositis, peri-implantitis

SUMMARY:
68 patients underwent the aMMP-8 chair-side test as well as clinical traditional measurement methods. Those who had one or more implants in their mouth were selected as patients. The condition of the attachment tissues of these implants is monitored at a control visit after five years.

DETAILED DESCRIPTION:
Patients who arrive for maintenance follow-up are included in the study. The trational measurement technique is used to follow the health of peri-implant tissues.

ELIGIBILITY:
Inclusion Criteria:

* the participation previously study implant patient

Exclusion Criteria:

* has not received antibiotic treatment within 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-11 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Tratitional measurement | 5 years
  the depth of the implant's gum pocket
Traditional measure | through study completion, an average of 5 year
  Bleedin on probing
Biomarker test | through study completion, an average of 5 year
  aMMP-8 tests, taking peri-implant sulcus fluid

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Study Director — University of Helsinki
Locations (1):
- Department of Oral and Maxillofacial Diseases, Head and Neck Center, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lahteenmaki H, Umeizudike KA, Heikkinen AM, Raisanen IT, Rathnayake N, Johannsen G, Tervahartiala T, Nwhator SO, Sorsa T. aMMP-8 Point-of-Care/Chairside Oral Fluid Technology as a Rapid, Non-Invasive Tool for Periodontitis and Peri-Implantitis Screening in a Medical Care Setting. Diagnostics (Basel). 2020 Aug 5;10(8):562. doi: 10.3390/diagnostics10080562. PMID 32764436
- [Background] Natto ZS, Almeganni N, Alnakeeb E, Bukhari Z, Jan R, Iacono VJ. Peri-Implantitis and Peri-Implant Mucositis Case Definitions in Dental Research: A Systematic Assessment. J Oral Implantol. 2019 Apr;45(2):127-131. doi: 10.1563/aaid-joi-D-18-00097. Epub 2018 Dec 17. PMID 30557088
- [Background] Sorsa T, Tervahartiala T, Leppilahti J, Hernandez M, Gamonal J, Tuomainen AM, Lauhio A, Pussinen PJ, Mantyla P. Collagenase-2 (MMP-8) as a point-of-care biomarker in periodontitis and cardiovascular diseases. Therapeutic response to non-antimicrobial properties of tetracyclines. Pharmacol Res. 2011 Feb;63(2):108-13. doi: 10.1016/j.phrs.2010.10.005. Epub 2010 Oct 16. PMID 20937384
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952